CLINICAL TRIAL: NCT06898645
Title: Clinical Study on the Effecacy of Transcranial Magnetic Stimulation of Intermittent Theta Pulse Stimulation(iTBS) Navigated Targeting the Cerebellum in the Treatment of Hereditary Spinocerebellar Ataxia
Brief Title: Efficacy of Cerebellar Transcranial Magnetic Stimulation to Treat Hereditary Spinocerebellar Ataxias
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20242432
Record Dates: First submitted 2025-02-04; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-01

CONDITIONS: Spinocerebellar Ataxias
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Intervention Model Description: randomly divided into intervention group and sham stimulation group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active stimulation (Experimental): navigated iTBS (Intermittent theta-burst stimulation) targeting the cerebellum
  Interventions: Device: navigated iTBS (Intermittent theta-burst stimulation) targeting the cerebellum
- sham stimulation (Sham Comparator): Sham stimulation was delivered via the built-in mode of the stimulator with 10% RMT intensity.
  Interventions: Device: navigated iTBS (Intermittent theta-burst stimulation) targeting the cerebellum

INTERVENTIONS:
Device: navigated iTBS (Intermittent theta-burst stimulation) targeting the cerebellum — 1,800 pulses per session for unilateral cerebellum, 50-minute intersession interval, 80% resting motor threshold, total 75600 pulse number.

SUMMARY:
Spinocerebellar ataxia (SCA) is a type of autosomal dominant ataxia and there is currently no effective treatment. The goal of this clinical trial is to learn the efficacy of navigated iTBS (Intermittent theta-burst stimulation) targeting the cerebellum to treat hereditary spinocerebellar ataxias in adults and explore the role and neural plasticity mechanisms. It will also learn about the safety of cerebellar transcranial magnetic stimulation. The main questions it aims to answer are:

1. Does navigated iTBS targeting the cerebellum improve the symptoms and clinical scale score of ataxias?
2. Safety evaluation measures included treatment-related dizziness, head and neck pain, tinnitus, hearing loss, and epilepsy. Adverse reactions were reported by both subjects and investigators.

Participants will:

1. Navigated iTBS targeting the cerebellum or sham stimulation every day for 7 day,
2. Assessments were made at baseline, within 24 hours after the end of treatment, after 12 weeks, and after 24 weeks of telephone follow-up.

DETAILED DESCRIPTION:
1. Gait analysis, electroencephalogram (EEG), functional magnetic resonance (fMRI) and a series of clinic scales were used to further observe the therapeutic effect and reveal the possible mechanism of neuroplasticity.
2. Forty-two iTBS sessions（1,800 pulses per session, 50-minute intersession interval） were delivered as 6 daily sessions over 7 consecutive days at 80% resting motor threshold (adjusted for cortical depth).

ELIGIBILITY:
Inclusion Criteria:

* SCA1/2/3 patients confirmed by genetic testing
* aged 18-65 years
* presence of ataxia with a score3-20 on the Scale for the Assessment and Rating of Ataxia (SARA) and a score<60 on the International Cooperative Ataxia Rating Scale (ICARS)
* Signed informed consent by patients or their family members

Exclusion Criteria:

* Patients with serious medical conditions (such as kidney failure, liver disease) and uncontrolled high blood pressure or diabetes
* Patients with severe cognitive and behavioral disorders or mental illness
* Pregnant and lactating patients; Use other ongoing clinical medications, except for neuroprotective agents such as coenzyme Q10, butylphthalein, or cyticholine; If patients are taking valproate, riluzole and other drugs but they and their guardians have a strong desire for treatment, they can be evaluated again after washout.
* History of stroke, encephalitis and epilepsy
* Pacemakers, electronic devices and intracranial metal objects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The change from baseline score on ICARS(International Cooperative Ataxia Rating Scale) | at baseline, within 24 hours after the end of treatment, after 12 weeks, and within 24 hours after the end of the second round of treatment
  International Cooperative Ataxia Rating Scale contains four subscales on a scale of 0 to 100, with higher scores indicating more severe ataxia

SECONDARY OUTCOMES:
The change from baseline score on SARA(Scale for the Assessment and Rating of Ataxia) | at baseline, within 24 hours after the end of treatment, after 12 weeks, and within 24 hours after the end of the second round of treatment
  Scale for the Assessment and Rating of Ataxia contains eight items on a scale of 0 to 40, with higher scores indicating more severe ataxia
Gait analysis | at baseline, within 24 hours after the end of treatment, after 12 weeks, and within 24 hours after the end of the second round of treatment
  The instrumented gait analysis showed that step width, step length
scalp electroencephalogram | at baseline, within 24 hours after the end of treatment, after 12 weeks, and within 24 hours after the end of the second round of treatment
  TMS combined with EEG
Safety evaluation measures | within 24 hours after the end of treatment
  Incidence and severity of side effects

OTHER OUTCOMES:
The change from baseline score on MMSE(Mini-mental state examination) | at baseline, within 24 hours after the end of treatment, after 12 weeks, and within 24 hours after the end of the second round of treatment
  Assesse cognitive function (orientation, memory, attention, calculation, language ability, etc.)
MOCA(Montreal Cognitive Scale) | at baseline, within 24 hours after the end of treatment, after 12 weeks, and within 24 hours after the end of the second round of treatment
  A rapid cognitive assessment tool designed to evaluate cognitive dysfunction, covering 11 assessment items across 8 cognitive domains: attention and concentration, executive function, memory, language, visuospatial skills, abstract thinking, calculation, and orientation.
HAMA(Hamilton anxiety scale) | at baseline, within 24 hours after the end of treatment, after 12 weeks, and within 24 hours after the end of the second round of treatment
  Assess the severity of anxiety symptoms in patients
HAMD(Hamilton depression scale) | at baseline, within 24 hours after the end of treatment, after 12 weeks, and within 24 hours after the end of the second round of treatment
  Assess the severity of depressive symptoms
PSQI(Pittsburgh sleep quality Index) | at baseline, within 24 hours after the end of treatment, after 12 weeks, and within 24 hours after the end of the second round of treatment
  A self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval
The 9-Hole Peg Test | at baseline, within 24 hours after the end of treatment, after 12 weeks, and within 24 hours after the end of the second round of treatment
  A common fine motor test used in occupational therapy assessments to collect a baseline on fine motor skills, dexterity, hand-eye coordination, motor planning, and more
10-m walking test | at baseline, within 24 hours after the end of treatment, after 12 weeks, and within 24 hours after the end of the second round of treatment
  The 10 Metre Walk Test is a performance measure used to assess walking or gait speed in meters per second over a short distance and can be employed to determine functional mobility, gait, and vestibular function